CLINICAL TRIAL: NCT06819761
Title: A Short, Open, Phase 0 Study to Demonstrate the Viability of the Lozenge Dosage Form to Deliver SALI-10 Oral Probiotics
Brief Title: Determining the Viability a Lozenge Dosage for Probiotics
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ostia Sciences (Industry)
Responsible Party: Principal Investigator, Michael Glogauer, Principal Investigator, Ostia Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: OstiaPhase0_2025_02Feb_04
Record Dates: First submitted 2025-02-04; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Delivery Systems; Oral Health
Keywords: Probiotics; Oral cavity; Lozenge; Dosage Forms

STUDY DESIGN:
Intervention Model Description: Open-label, single-arm, exploratory pilot study to be completed over 7 days with 8-10 participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Receives Probiotic Lozenge (Experimental): This study is an open-label, single-arm, exploratory pilot study to be completed over 7 days with 8-10 participants. Participants will self-administer one lozenge containing S. salivarius SALI-10 (10 billion CFU/lozenge) each night after brushing and before bed. Every participant will be given 7 SALI-10 lozenges.
  1. The aim of this study is to determine the short-term ability of the Streptococcus salivarius SALI-10 lozenges delivery system to modify the human oral microbiome composition and Oral Inflammatory Load (OIL). Specifically, we aim to:
     * Assess the change in salivary levels of periodontal-disease-associated bacteria (e.g., P. gingivalis, T. forsythia, T. denticola, and P. micra).
     * Determine the change in beneficial bacteria levels (e.g., S. salivarius, S. parasanguinis).
     * Evaluate the change in Oral Inflammatory Load (OIL) by measuring oral neutrophil counts.
  2. To monitor the short-term adherence of the 8-10 participants to the clinical protocol.
  Interventions: Dietary Supplement: Salivarius SALI-10

INTERVENTIONS:
Dietary Supplement: Salivarius SALI-10 — Lozenge with 10B CFU (Colony Forming Units)

SUMMARY:
Gingivitis is an oral disease condition affecting 50% to 90% of adults globally. Gingivitis is a reversible inflammatory condition caused by the accumulation of dental plaque and the associated disruption of the host-microbial homeostasis. During gingivitis, the microbial community shifts from gram-positive health-associated bacteria, to gram-negative disease associated species. This shift triggers inflammatory responses, leading to tissue damage and, in some cases, progression to periodontitis.

A promise area of oral health is treating the oral cavity with gram-positive probiotics to improve oral health. One promising candidate is S. salivarius SALI-10. Typically oral probiotics are dosed to the oral cavity using lozenges. This study is a pre-clinical Phase 0 trial to determine is a lozenge is a viable dosage form for the delivery of salivarius SALI-10 oral probiotics.

DETAILED DESCRIPTION:
Gingivitis is an oral disease condition affecting 50% to 90% of adults globally (Albandar and Rams, 2002). The gingivitis pathology can be reversed by reduction or removal of microbial plaque that accumulates on hard and soft tissues and is considered standard of care in the industry (Berezow Alex and Darveau Richard, 2010, van der Weijden and Slot, 2011). Regular oral hygiene in combination with therapeutics that delivers an anti-microbial benefit is thought to mitigate the onset of gingivitis (van der Weijden and Slot, 2011, Gunsolley, 2006). However, testing therapeutics for prophylaxis benefit to mitigate development of gingivitis has not been fully examined.

Neutrophils, a type of white blood cell (leukocyte), represent a key component of the innate defence system that protects periodontal tissue from both gingivitis and periodontitis. Not only are they the first line of cellular defence, but they are among the most abundant leukocytes within the periodontal tissues (Hirschfeld, 2020). For example, gingivitis is associated with a significant increase in the number of neutrophils that migrate to periodontal tissue. In contrast, individuals with too few neutrophils brought about by either congenital deficiencies in neutrophil numbers, or transit (LAD 1 and 2) or have an induced neutropenia by chemical induction with antimitotic agents such as cyclophosamide invariably develop periodontitis. Likewise, studies in KO mice that are defective in neutrophil transit also develop periodontitis. Consistent with the key contribution of neutrophils to both gingivitis and periodontitis, neutrophil transit to gingival tissue is highly regulated. The periodontium contains a highly orchestrated expression of select innate host defense mediators that facilitate the transit of neutrophils from the highly vascularized gingival tissue to the gingival crevice, where they form a "wall" between the host tissue and the dental plaque biofilm.

Gingivitis is a reversible inflammatory condition caused by the accumulation of dental plaque and the associated disruption of the host-microbial homeostasis. During gingivitis, the microbial community transitions from being dominated by gram-positive health-associated bacteria, such as Streptococcus species, to gram-negative periopathogens, including species of the genera Porphyromonas, Tannerella, Treponema and Prevotella. This dysbiotic shift triggers inflammatory responses, leading to tissue damage and, in some cases, progression to periodontitis.

A recent study (Kerns, 2023) on human experimental gingivitis identified three distinct host response phenotypes-high, low, and slow responders-based on clinical, inflammatory, and microbial parameters:

1. High Responders: Rapid plaque accumulation accompanied by a significant increase in gram-negative periopathogens and elevated inflammatory markers, such as interleukin-1β (IL-1β).
2. Low Responders: Similar plaque accumulation to high responders but lower inflammation, suggesting a more muted host response to bacterial dysbiosis.
3. Slow Responders: Delayed plaque accumulation and microbial succession, with prolonged dominance of health-associated Streptococcus species. This group exhibited delayed or reduced inflammation, demonstrating a more resilient microbial community and host response.

The microbial analysis revealed that the persistence of beneficial Streptococcus species, such as S. sanguinis and S. oralis, in slow and low responders correlates with a protective effect against the emergence of periopathogens and the associated inflammatory cascade. Conversely, the loss of these beneficial bacteria in high responders was linked to more severe inflammation, highlighting the critical role of the oral microbiome in modulating gingivitis severity.

Lantibiotic salivaricins are polycyclic peptides containing lanthionine and/or β-methyllanthionine residues that are produced by certain strains of Streptococcus salivarius, which almost exclusively reside in the human oral cavity. These molecules importance stems from their antimicrobial activity towards relevant oral pathogens which has been applied through the development of salivaricin-producing probiotic strains. However, salivaricins may also prove to be of great value in the development of new and novel antibacterial therapies in this era of emerging antibiotic resistance (Barbour, Wescombe, & Smith, 2020). In a study by Barbour & Philip 2014, they found that the bacteriocin, levan-sucrase production and basic safety features of S. salivarius strains isolated from healthy Malaysian subjects demonstrating their potential for use as probiotics. A new bacteriocin production medium was developed with potential scale up application for pharmaceuticals and probiotics from S. salivarius generating different lantibiotics. This is relevant for the clinical management of oral cavity and upper respiratory tract in the human population. Appendix 1 includes a summary table that lists the relevant clinical trials that utilized S. salivarius.

Proposed Solution: S. salivarius SALI-10

We propose using a novel strain, Streptococcus salivarius SALI-10, as a targeted microbial intervention to modulate the oral microbiome and prevent gingivitis. S. salivarius SALI-10 is hypothezised to:

* Maintain a stable population of beneficial streptococci during plaque accumulation.
* Inhibit the growth of periopathogens such as Porphyromonas, Tannerella and Prevotella through competition and production of Salivaricin 10.
* Delay or suppress the dysbiotic shift to gram-negative dominance, thereby reducing the inflammatory response.

By preserving microbial homeostasis, SALI-10 may emulate the microbial resilience observed in slow responders, offering a novel strategy for gingivitis prevention.

Before the therapeutic value of Streptococcus salivarius SALI-10 can be assessed, its dosage form must be validated. The classical method of delivering oral probiotics is in a lozenge form, having the individual suck on the lozenge until it dissolves. Once it is verified that this dosage form works for Streptococcus salivarius SALI-10, a full clinical trial to determine its therapeutic viability can be conducted.

2. STUDY OJECTIVES

1. The aim of this study is to determine the short-term ability of the Streptococcus salivarius SALI-10 lozenges delivery system to modify the human oral microbiome composition and Oral Inflammatory Load (OIL). Specifically, we aim to:

   * Assess the change in salivary levels of periodontal-disease-associated bacteria (e.g., P. gingivalis, T. forsythia, T. denticola, and P. micra).
   * Determine the change in beneficial bacteria levels (e.g., S. salivarius, S. parasanguinis).
   * Evaluate the change in Oral Inflammatory Load (OIL) by measuring oral neutrophil counts.
2. To monitor the short-term adherence of the 8-10 participants to the clinical protocol

3. STUDY OVERVIEW

This study is designed as an open-label, single-arm, exploratory pilot study to be completed over 7 days with 8-10 participants. Participants will self-administer one lozenge containing S. salivarius SALI-10 (10 billion CFU/lozenge) each night after brushing and before bed. Participants will complete two (2) home sample kits, one before and one after the 7 days.

5. TEST PRODUCTS/INTERVENTIONS Each participant will receive seven (7) mint-flavoured SALI-10 lozenges. They will be instructed to take a lozenge daily after brushing by letting it dissolve in the mouth. The participants will be using the SALI-10 lozenges throughout the study. Each participant will also receive four (4) home administered test kits: two (2) Saliva Collection Kits, and two (2) Saline Rinse Collection Kits.

5.2 Dispensing, Storage, and Accountability Once pre-screened, all participants will receive all study materials in the mail. This will include the seven (7) lozenges, and the four (4) home administered test kits: two (2) Saliva Collection Kits, and two (2) Saline Rinse Collection Kits. The subjects will follow provided instructions on when and how to brush their teeth. These instructions are explained in the procedure section.

The test kits are self-contained commercially available kits that include all instructions of use. Participants will be provided instructions on how drop off the samples to Ostia Sciences Inc at 124 Edward St., Toronto, Suit 463, ON Canada M5G 1G6.

Participants will be instructed to throw out all study materials that the end of the 7-day trial.

6. STUDY PROCEDURES

6.2 Product Dispensing and Use at Home

The product will be mailed to the participant in a sealed box that will include instructions for at-home use and safety information, including emergency contact details. To monitor patient compliance, clinical study manager will request an email confirmation at the end of the trial that all 7 lozenges were consumed. Subjects will be assigned a unique identification number in chronological order (e.g., from 1 to 10) as they enroll in the study. Subjects will be instructed to avoid using any other oral hygiene products. There will be no dietary restrictions during the study.

Subjects will be instructed to brush their teeth twice daily (morning and evening) for two minutes each time with a toothpaste and toothbrush and floss.

The SALI-10 lozenges will be pre-packed when given to each participant.

6.3 Telephone Pre-Screening Potential study participants who contact the clinical trial coordinator for more information about the study via email will then be contacted via telephone. At this stage the Recruitment Questionnaire (Appendix 3) will be completed to determine whether they are eligible for the screening phase of the study. If the subject is deemed eligible they will be given the Informed Consent Form to read and ask any questions they may have and sign. The screening will be carried out until ten (10) subjects are enrolled.

There will no in-person visits. Study participants will be mailed all study materials, which included the seven (7) lozenges, and the four (4) home administered test kits: two (2) Saliva Collection Kits, and two (2) Saline Rinse Collection Kits. Subjects will also receive the study product for use at home with directions.

6.5 Day 0 (Baseline)

Participants will utilize one (1) Saliva Collection Kit, and one (1) Saline Rinse Collection Kit. They will drop off the samples to Ostia Sciences as per the given instructions. After sample collection, participants will begin using the lozenges daily for 7 days. The participants will take one lozenge after brushing. They will allow the lozenges to dissolve without biting or swallowing and avoid eating and drinking for one hour. The participants will be instructed on proper oral hygiene and will be instructed to continue their home oral hygiene in addition to use of their assigned product for 7 days (1 week). The participants will be instructed to discard the lozenges' container at the end of the study.

6.6 Day 7 (Completion)

24 hours after using the seventh (7th) lozenge, participants will utilize one (1) Saliva Collection Kit, and one (1) Saline Rinse Collection Kit. They will drop off the samples to Ostia Sciences as per the given instructions. Study participants will discard any remaining study materials they may have. Through email, the study manager will confirm adherence to protocol and provide post-study instructions. The subjects will be informed that this is the end of the study. They will be told that they may resume their regular oral hygiene. Afterwards, we will ask the participants for their feedback in regards to their experience.

7. STUDY PROCEDURES AND CLINICAL REGISTRATIONS

7.7 Saliva and Oral Rinse Samples

The Saliva Collection Kit is the SuperSAL2 Universal Saliva Collection Kit, Instructions are found in Appendix 10. The saliva samples will be processed and will be analyzed by DNA

DNA extraction, then qPCR will be used to quantify the full change of specific bacteria in the saliva samples, specifically pathogenic bacteria (P. gingivalis, T. forsythia, T. denticola, P. micra) and beneficial bacteria (S. salivarius, S. parasanguinis).

The Oral Rinse Collection Kit is produced by Ostia Sciences, with instructions found in Appendix 11. There Oral rinse samples will be analyzed for oral neutrophil counts as a marker of Oral Inflammatory Load (OIL).

Since all research projects will be done on de-identified samples, it will not be possible to return individual results to participants. All samples will be destroyed immediately after testing. Because all research will be done on de-identified, aggregated data, it will not be possible to withdraw the data from a specific participant when samples are withdrawn from the study.

8.0 STATISICAL ANALYSES

For statistical analysis, full change of the microbes and the OIL will be compared between Baseline and Day 7 Completion using paired Wilcoxon test.

9.0 REPORT OF ADVERSE EVENTS

Subjects will be told of any possible adverse reactions or side effects from exposure to this method or product. Oral irritation is possible. If side effects occur, it is expected to be mild and temporary. Any event will stop when the subject stops being exposed to the instrument or returns to their normal oral hygiene. The investigators will record any and all adverse reactions and report this documentation to the Product Safety Assurance Department. The nature of the reaction and any correlation with product usage will be assessed. If the evidence indicates that the adverse reaction may be due to product usage, the subject will be instructed to discontinue product use and appropriate treatment will be provided. In the event of an adverse experience, emergency or other problems or questions regarding your participation in this study you can contact the following investigators:

Dr. Michael Glogauer at (905) 973-0664. In the event of a medical emergency, please contact your physician.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female volunteers aged 18-70 years
2. In good general health, ASA I
3. Non-smokers
4. Fluent in English

Exclusion Criteria:

1. Presence of orthodontic bands.
2. Presence of partial removal dentures.
3. Dental pain at time of screening.
4. History of allergy to a consumer or personal care products or dentifrice ingredients as determined by the dental profession monitoring the study.
5. Participation in any other clinical study or test panel within one month before entering the study.
6. Current use of anti-inflammatory, antibiotics, or antimicrobial drugs or within the last 30 days of enrolment.
7. History of periodontal disease.
8. History of systemic inflammatory or immune conditions
9. Pregnant or nursing women.
10. Use of tobacco products.
11. Long-term antibiotic or anti-inflammatory therapy.
12. Medical condition or any current usage of medication that the investigator considers may compromise the subject's safety as well as the quality of the study results;
13. Use of any concomitant medication.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Changes in microbiome composition in the oral cavity | From enrollment to the end of treatment at 7 days
  * Assess the change in salivary levels of periodontal-disease-associated bacteria (e.g., P. gingivalis, T. forsythia, T. denticola, and P. micra).
  * Determine the change in beneficial bacteria levels (e.g., S. salivarius, S. parasanguinis).

SECONDARY OUTCOMES:
Oral Inflammatory Load | From enrollment to the end of treatment at 7 days.
  Evaluate the change in Oral Inflammatory Load (OIL) by measuring oral neutrophil counts.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Glogauger, MD, Principal Investigator — Ostia Sciences Inc
Locations (1):
- Ostia Sciences Inc, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
This is a Phase 0 trial, and no individual participant data will be kept.

REFERENCES:
- [Background] Wellappuli NC, Fine N, Lawrence HP, Goldberg M, Tenenbaum HC, Glogauer M. Oral and Blood Neutrophil Activation States during Experimental Gingivitis. JDR Clin Trans Res. 2018 Jan;3(1):65-75. doi: 10.1177/2380084417742120. Epub 2017 Nov 20. PMID 30938653
- [Background] van der Weijden F, Slot DE. Oral hygiene in the prevention of periodontal diseases: the evidence. Periodontol 2000. 2011 Feb;55(1):104-23. doi: 10.1111/j.1600-0757.2009.00337.x. No abstract available. PMID 21134231
- [Background] LOE H, THEILADE E, JENSEN SB. EXPERIMENTAL GINGIVITIS IN MAN. J Periodontol (1930). 1965 May-Jun;36:177-87. doi: 10.1902/jop.1965.36.3.177. No abstract available. PMID 14296927
- [Background] Kerns KA, Bamashmous S, Hendrickson EL, Kotsakis GA, Leroux BG, Daubert DD, Roberts FA, Chen D, Trivedi HM, Darveau RP, McLean JS. Localized microbially induced inflammation influences distant healthy tissues in the human oral cavity. Proc Natl Acad Sci U S A. 2023 Oct 10;120(41):e2306020120. doi: 10.1073/pnas.2306020120. Epub 2023 Oct 2. PMID 37782795
- [Background] Gunsolley JC. A meta-analysis of six-month studies of antiplaque and antigingivitis agents. J Am Dent Assoc. 2006 Dec;137(12):1649-57. doi: 10.14219/jada.archive.2006.0110. PMID 17138709
- [Background] Gallagher H, Ramsay SC, Barnes J, Maggs J, Cassidy N, Ketheesan N. Neutrophil labeling with [(99m)Tc]-technetium stannous colloid is complement receptor 3-mediated and increases the neutrophil priming response to lipopolysaccharide. Nucl Med Biol. 2006 Apr;33(3):433-9. doi: 10.1016/j.nucmedbio.2005.12.014. Epub 2006 Mar 9. PMID 16631093
- [Background] Berezow AB, Darveau RP. Microbial shift and periodontitis. Periodontol 2000. 2011 Feb;55(1):36-47. doi: 10.1111/j.1600-0757.2010.00350.x. No abstract available. PMID 21134227
- [Background] Barbour A, Wescombe P, Smith L. Evolution of Lantibiotic Salivaricins: New Weapons to Fight Infectious Diseases. Trends Microbiol. 2020 Jul;28(7):578-593. doi: 10.1016/j.tim.2020.03.001. Epub 2020 Apr 6. PMID 32544444
- [Background] Barbour A, Philip K. Variable characteristics of bacteriocin-producing Streptococcus salivarius strains isolated from Malaysian subjects. PLoS One. 2014 Jun 18;9(6):e100541. doi: 10.1371/journal.pone.0100541. eCollection 2014. PMID 24941127
- [Background] Albandar JM, Rams TE. Global epidemiology of periodontal diseases: an overview. Periodontol 2000. 2002;29:7-10. doi: 10.1034/j.1600-0757.2002.290101.x. No abstract available. PMID 12102700